CLINICAL TRIAL: NCT00002114
Title: A Double-Blind, Randomized Parallel Group Study Comparing Procysteine to Placebo in HIV-Infected Patients Who Are Taking Antiretroviral Nucleosides
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Free Radical Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 215A; CN9202D
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1994-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — 2-oxothiazolidine-4-carboxylic acid

INTERVENTIONS:
Drug: Procysteine

SUMMARY:
To compare the efficacy and safety of orally administered Procysteine with placebo in HIV-infected patients who are receiving 1 of the following: (1) zidovudine (AZT) alone; (2) didanosine (ddI) alone; (3) AZT plus ddI; or (4) AZT plus zalcitabine (ddC).

DETAILED DESCRIPTION:
All patients must receive treatment with antiretroviral nucleosides in addition to study treatment. Patients are randomized equally into 1 of 3 outpatient dosage groups. Group 1 receives placebo; Group 2 receives a low dose of Procysteine; and Group 3 receives a higher dose of Procysteine. Patients receive study treatment for 6 months (total duration of patient participation is 30 weeks).

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

Antiretroviral nucleosides (AZT alone, ddI alone, AZT plus ddI, or AZT plus ddC). Regimen may be altered on or after Week 16.

Allowed:

* Appropriate topical treatment or local radiotherapy for KS.
* Treatment or prophylaxis for opportunistic infections, including pentamidine, cotrimoxazole, acyclovir, fluconazole, etc., at the discretion of the investigator.

Patients must have:

* Documented serologic evidence confirming HIV infection.
* Ability to participate in an outpatient study for at least 26 weeks.
* Either:
* (a) diagnosis of AIDS or AIDS-Related Complex (ARC) with CD4 count of 50 - 300 cells/mm3, or (b) CD4 count of 50 - 200 cells/mm3 and no symptoms of AIDS (asymptomatic). (Note:
* Patients whose AIDS-defining condition is Kaposi's sarcoma alone must have CD4 count of 50 - 200 cells/mm3.)

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Evidence of organ involvement with CMV and/or positive blood cultures for Mycobacterium avium.
* Life expectancy less than 26 weeks.
* Malignancy or advancing Kaposi's sarcoma (KS) with advancing or unstable skin lesion, or known or suspected visceral disease which requires systemic cytotoxic, myelosuppressive chemotherapy.
* Stage 2 or greater AIDS-dementia complex (ADC), defined as ability to perform basic activities of self-care but inability to work or maintain more demanding aspects of daily life as a result of an acquired decrease in cognitive CNS-related motor function characteristic of ADC.
* Psychological or emotional problems that prevent adequate compliance with study therapy.

Concurrent Medication:

Excluded:

* Daily Vitamin C dosage greater than 1,000 mg or daily Vitamin E dosage greater than 100 units.
* N-acetylcysteine, cysteine, or glutathione.
* Any investigational drug.
* Systemic chemotherapy.

Patients with the following prior conditions are excluded:

* History of organ involvement with cytomegalovirus (CMV) and/or positive blood cultures for Mycobacterium avium.
* Intractable diarrhea, defined as greater than 4 bowel movements per day for at least 2 weeks.
* History of seizures which have not been controlled with appropriate anticonvulsant medications within the previous 6 months.

Prior Medication:

Excluded:

* Any investigational agent or biological response modifier (including interferon or corticosteroids) within 1 month of study entry.
* Use of erythropoietin (EPO), G-CSF, or GM-CSF within 28 days of randomization.

Risk Behavior:

Excluded:

Active alcohol or drug abuse.

Required:

Antiretroviral nucleosides (AZT alone, ddI alone, AZT plus ddI, or AZT plus ddC) for at least 3 months prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125
Dates: Study Completion 1994-01